CLINICAL TRIAL: NCT05339204
Title: Prospective Multicenter Randomized Controlled Clinical Trial for Evaluation the Role of Allo-HSCT in the First Complete Remission, MRD-negative After the First Course, in Patients With AML Under the Age of 60 Years
Brief Title: The Role of Allo-HSCT in MRD-negative Patients With AML Under the Age of 60 Years in the First Complete Remission
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Research Center for Hematology, Russia (Network)
Collaborators: Botkin Hospital (Other); St. Petersburg State Pavlov Medical University (Other); Federal State Budgetary Institution, V. A. Almazov Federal North-West Medical Research Centre, of the Ministry of Health (Other); Federal Research Clinical Center of Federal Medical & Biological Agency, Russia (Other Government); Regional Clinical Hospital of Yaroslavl (Unknown); Nizhny Novgorod regional clinical hospital named after N.A.Semashko (Unknown); Clinical hospital №1 of Sverdlovsk region (Unknown); Irkutsk regional clinical hospital, winner of the "Mark of the Honor" award (Unknown); The Federal State-Financed Scientific Institution Kirov Research Institute of Hematology and Blood T (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AML-21
Record Dates: First submitted 2022-04-14; First posted 2022-04-21 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: AML
Keywords: AML, MRD, allo-HSCT, CR1, adult
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- allo-HSCT (Experimental): Patients with AML in CR1, MRD-negative after first course recieve allo-HSCT
  Interventions: Procedure: allo-HSCT
- Chemo (Active Comparator): Patients with AML in CR1, MRD-negative after first course continue chemotherapy
  Interventions: Procedure: allo-HSCT

INTERVENTIONS:
Procedure: allo-HSCT — allo-HSCT from any type of donor

SUMMARY:
Depending on the variant of the disease, patients are divided into 3 groups: A, B and C. Group A include patients with acute myeloid leukemia (AML) inv(16)(p13.1q22) or t(16;16)(p13.1;q22); CBFB-MYH11, group B - AML with t(8;21)(q22;q22.1); RUNX1-RUNX1T1, AML with normal karyotype with or without gene mutations (FLT3, NPM1, CEBPa) regardless of the allele ratio, and also AML with cytogenetic abnormalities not classified as those within groups A/C, group C - AML with myelodysplasia-related changes. Patients from group A receive treatment according to the scheme: 2 courses "7+3", 2 courses "FLAG", then - 6 courses of maintenance therapy according to the scheme "5+5". Patients from group B are given one course of "7+3". After that, their minimal residual disease (MRD) status is assessed. In case MRD negativity is achieved after the 1st course of "7 +3", randomization is carried out: branch 1 - therapy is similar to therapy for patients from group A (4 courses of induction and consolidation + 6 courses of maintenance chemotherapy (CT), allogeneic hematopoietic stem cell transplantation (allo-HSCT) is not planned), branch 2 - performing allo-HSCT should be done as soon as possible (before the start of maintenance CT is most desirable). If MRD negativity is not achieved after the 1st course of "7+3", the patient is given CT according to the standard program, followed by mandatory allo-HSCT. Patients from group C are treated either according to the "Aza-Ida-Ara-C" scheme, or according to the "Ven-DAC /AZA" scheme, followed by mandatory allo-HSCT.

DETAILED DESCRIPTION:
"7+3" regimen:

1. Cytarabine 200 mg/m2 (IV continuous infusion over 24 hours), days 1-7
2. Daunorubicin 60 mg/m2 (IV bolus), days 1-3

"FLAG" regimen:

1. Fludarabine 25 mg/m2 (IV in 30 minutes), days 1-5
2. Cytarabine 1500 mg/m2 (IV in 3 hours), days 1-5
3. Granulocyte colony-stimulating factor 5 mcg/kg (subcutaneous injection), from day 6 until regression of cytopenia

"Aza-Ida-Ara-C" regimen:

1. Azacitidine 75 mg/m2 (subcutaneous injection), days 1-3
2. Idarubicin 3 mg/m2 (IV bolus), days 4-10
3. Cytarabine 15 mg/m2 twice a day (subcutaneous injection), days 4-17

"Ven-DAC/AZA"

1. Venetoclax 400 mg once daily (PO), days 1-28
2. Either Azacitidine or Decitabine Azacitidine 75 mg/m2 (subcutaneous injection), days 1-7 Decitabine 20 mg/m2 (IV in 60 minutes). days 1-5

"5+5" regimen

1. Cytarabine 50 mg/m2 twice a day (subcutaneous injection), days 1-5
2. Mercaptopurine 30 mg/m2 twice a day (PO), days 1-5

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed, previously untreated AML;
2. Age from 18 to 59 years;
3. Somatic status - ECOG < 3.

Exclusion Criteria:

1. previous chemotherapy for AML;
2. pregnancy;
3. relapses and refractory forms of AML;
4. acute promyelocytic leukemia;
5. blast crisis of chronic myeloid leukemia;
6. de novo AML with t(9;22);
7. AML transformed from MDS or MPN after treatment, for which a different protocol is provided;
8. Blastoid plasmacytoid dendritic cell neoplasia (with the exception of cases when a small population of plasmacytoid dendritic progenitors is detected in the leukemic neoplasia).
9. Undifferentiated acute leukemia

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival for AML in CR1 with MRD-negativity after first course of chemo | 5 years
Relapse probability | 5 years

SECONDARY OUTCOMES:
Overall survival | 5 years
Disease-free survival | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- National Research Center for Hematology, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Yes